CLINICAL TRIAL: NCT00639652
Title: Observational Study: Recurrence Rate and Esthetic Outcome After Excision of Basal Cell Carcinomas Excluded From Trial NCT00515970
Brief Title: Recurrence Rate and Esthetic Outcome After Excision of Basal Cell Carcinomas Excluded From Trial NCT00515970
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Helmut Breuninger, Department of Dermatology, Eberhard Karls University
Other Study IDs: 16/2008BO2
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2008-03

CONDITIONS: Carcinoma, Basal Cell
Keywords: Carcinoma, Basal Cell; 3D-histology; Micrographic surgery; Mohs surgery; Shave excision; Recurrence; Esthetic outcome
MeSH Terms: conditions — Carcinoma, Basal Cell; Recurrence | interventions — Mohs Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Paraffinized histology blocks and sections.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. 3D-histology: Nodular, micronodular, or sclerosing BCCs
  Interventions: Procedure: 3D-histology
- 2. Shave excision: Superficial BCCs
  Interventions: Procedure: Shave excision

INTERVENTIONS:
Procedure: 3D-histology — The tumor is marked at the 12 o'clock-position. Excision with a safety margin between 2 and 10 mm, depending on tumor size and location. Plastic reconstruction. Removal of the specimen's margins and base as thin layers, using a scalpel. These primarily three-dimensional layers of the specimen's borders are flattened to one level and microscopically screened for tumor cells. 3D-histology is combined with representative vertical sections for histologic diagnosis. Consecutive excisions are performed topographically at the tumor-positive areas and 3D-histology is repeated until tumor-free margins are obtained.
  Other Names: Micrographic surgery; Histographic surgery; Mohs surgery
  Groups: 1. 3D-histology
Procedure: Shave excision — Tumor removal by shave excision with a safety margin. Healing by secondary intention. Histologic diagnosis of BCC type (nodular, superficial, morpheaform, micronodular, other type, mixed type) or diagnosis of another tumor than BCC. Comment on complete removal (R0 versus R1).
  Groups: 2. Shave excision

SUMMARY:
Currently, we conduct a prospective, randomized trial comparing the outcome of surgical excision with the outcome of curettage in nodular and superficial BCCs. Larger BCCs and micronodular or sclerosing BCCs are not included in the randomized study. They are mainly operated using three-dimensional histology (3D-histology, micrographic surgery). In this observational study we measure the cosmetic result and the recurrence rate of all BCCs not included in the randomized trial.

DETAILED DESCRIPTION:
1. Disinfection
2. Local anesthesia
3. Surgery
4. Dressing
5. Preparation with paraffin for histopathologic evaluation
6. Staining with hematoxylin-eosin
7. Adjuvant radiotherapy is not applied in any of our patients.
8. If histopathology discovers another tumor than BCC, the tumor is excluded.
9. If recurrence is suspected, a punch biopsy is taken. If recurrence is confirmed, the endpoint is achieved.
10. Patients who provide no feedback receive phone calls.
11. The patient receives a letter containing a list of the BCCs treated within the study. She or he is asked to visit the private practitioner with the list after 12 and 48 months (+/- 30 days) referring to the last operation in the recruitment period. The practitioner or the patient return the questionnaire to our department.
12. The letter contains a questionnaire about suspicion of recurrence of BCC.
13. The patient is asked to assess the esthetic outcome on a scale of excellent, good, satisfactory, mediocre, and poor.
14. The physician is asked to assess the esthetic outcome on a scale of excellent, good, satisfactory, mediocre, and poor.
15. When follow-up is closed for an individual patient, the reason is recorded:

    1. Planned end of follow-up after 48 months
    2. Patient has moved.
    3. Death (date of death)
    4. Consent withdrawn
    5. Meanwhile, the patient has become so ill or high-maintenance that no more follow-up visits can be planned.
    6. Recurrence of all of the patient's BCCs with histopathologic confirmation.

ELIGIBILITY:
Inclusion Criteria:

* BCCs excluded from the randomized trial NCT00515970

Exclusion Criteria:

* Treatment other than with 3D-histology or shave excision (e.g. deep surgical excision without 3D-histology)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: BCCs excluded from the randomized trial NCT00515970
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2007-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of basal cell carcinoma (BCC) | Within 4 years after surgery

SECONDARY OUTCOMES:
Subjective assessment of the esthetic outcome of the scar on a scale of excellent, good, satisfying, moderate, unfavorable; done by a private practitioner. | 12 and 48 months after surgery
Subjective assessment of the esthetic outcome of the scar on a scale of excellent, good, satisfying, moderate, unfavorable; done by the patient. | 12 and 48 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Breuninger, M.D., Study Chair — Eberhard Karls University Tuebingen, Department of Dermatology; Kay Brantsch, M.D., Principal Investigator — Eberhard Karls University Tuebingen, Department of Dermatology
Locations (1):
- Eberhard Karls University, Department of Dermatology, Tübingen, Germany